CLINICAL TRIAL: NCT01913119
Title: A Pilot Study of Romidepsin in Relapsed or Refractory Extranodal NK/T-cell
Brief Title: A Pilot Study of Romidepsin in Relapsed or Refractory Extranodal NK/T-cell Lymphoma
Acronym: Ro-ENKTL
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Principal Investigator, Won Seog Kim, professor, Samsung Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-10-059
Record Dates: First submitted 2013-07-19; First posted 2013-07-31 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Histologically Proven Extranodal NKTcell Lymphoma
Keywords: extranodal NKTcell lymphoma
MeSH Terms: interventions — romidepsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Romidepsin (Experimental): Day 1, 8, and 15 of a 28-day cycle Romidepsin Treatment is repeated until documented disease progression or unacceptable toxicity.
  Dose and administration: 4-hour infusion of 14 mg/m2
  Interventions: Drug: Romidepsin

INTERVENTIONS:
Drug: Romidepsin — Day 1, 8, and 15 of a 28-day cycle Romidepsin Treatment is repeated until documented disease progression or unacceptable toxicity.
  Dose and administration: 4-hour infusion of 14 mg/m2
  Other Names: Istodax

SUMMARY:
Extranodal NK/T-cell lymphoma is a rare disease entity with aggressive clinical course and poor prognosis. Currently, there is no treatment option for relapsed or refractory extranodal NK/T-cell lymphoma. Romidepsin is a histone deacetylase inhibitor which was approved for cutaneous T-cell lymphoma. A recent phase II study of romidepsin for relapsed/refractory peripheral T-cell lymphoma reported an overall response rate of 38% (95% confidence interval 24%-53%). The median duration of overall response was 8.9 months. Considering the median number of previous treatments in these patients was three (range 1-11), romidepsin has single agent activity against relapsed/refractory T-cell lymphoma. Thus, if the single agent activity of romidepsin is demonstrated, it could be a therapeutic agent for combination with salvage treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patient should belong to any one of following clinical situations

   1. Relapsed after salvage chemotherapy
   2. Relapsed after autologous stem cell transplantation
   3. Refractory to salvage chemotherapy or autologous stem cell transplantation
2. Adequate organ function as defined by the following criteria:

   1. Serum aspartate transaminase (AST; serum glutamic oxaloacetic transaminase (SGOT)) and serum alanine transaminase (ALT; serum glutamic pyruvic transaminase (SGPT)) ≤2.5 x local laboratory upper limit of normal (ULN), or AST and ALT less than or equal to 5 x ULN if liver function abnormalities are due to underlying malignancy
   2. Total serum bilirubin ≤ 1.5 x ULN
   3. Absolute neutrophil count (ANC) ≥1500/µL
   4. Platelets ≥ 75,000/µL
   5. Hemoglobin ≥ 9.0 g/dL (may be transfused or erythropoietin treated)
   6. Serum calcium ≤ 12.0 mg/dL
   7. Serum creatinine ≤ 1.5 x ULN
3. At least one measurable lesion
4. ECOG PS 0-2
5. Written informed consent
6. Over 20 years and under 80 years of age

Exclusion Criteria:

1. Previously received allogeneic stem cell transplantation
2. History of or known carcinomatous meningitis, or evidence of symptomatic leptomeningeal disease or secondary CNS involvement on CT or MRI scan.
3. Ongoing cardiac dysrhythmias of NCI CTCAE grade ≥2.
4. Pregnancy or breastfeeding.
5. Any Known cardiac abnormalities
6. HBV carrier
7. Positive for HIV

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Rate of overall disease control including CR, PR, and SD | Time between the date of treatment start and the date of death
  Overall rate of disease control including CR, PR and SD Overall survival: Time between the date of treatment start and the date of death due to any cause

SECONDARY OUTCOMES:
Number of participants with adverse events | from the date of informed consent signature to 30 days after last drug administration
  Number of participants with adverse events
Time to progression | from the date of first drug administration until the date of first documented progression
  Performing Cervical, Chest, Abdomen and Pelvis CT scan for the assessment
overall survival | from the date of first drug administration until the date of death
  Overall Survival will be measured from the date of first drug administration to the date of death from any cause.

CONTACTS AND LOCATIONS:
Locations (4):
- South Korea (4):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Korea Cancer Center Hospital, Nowon-gu, Seoul
  - Severance Hospital, Seodaemun-gu, Seoul
  - Asan Medical Center, Songpa-gu, Seoul